CLINICAL TRIAL: NCT05763420
Title: Clinical Efficacy of AH Plus Bioceramic Sealer in Root Canal Treatment of Molar Teeth: A Randomized Controlled Trial
Brief Title: Clinical Efficacy of AH Plus Bioceramic Sealer
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Ministry of Health, Kuwait (Other Government)
Collaborators: Kuwait Institute for Medical Specialization (Other Government)
Responsible Party: Principal Investigator, Ahmed Aldowaisan, Principal Investigator, Specialist in Endodontics, Ministry of Health, Kuwait
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2291
Record Dates: First submitted 2023-02-27; First posted 2023-03-10 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Root Canal Infection; Periapical Periodontitis; Periapical Diseases
MeSH Terms: conditions — Periapical Periodontitis; Periapical Diseases

STUDY DESIGN:
Intervention Model Description: Permuted block randomization using a block size of 4 will be used to randomly select 136 participants (68 participants in each group). The Study Randomizer website (http://www.studyrandomizer.com) will be utilized to generate the randomization list and participants will be assigned to the selected treatment group accordingly.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Participants will be blinded to the type of treatment they will receive to reduce bias in the reporting of pain.
  Since it is not possible to blind the care providers, they will only be informed of the type of treatment once cleaning and shaping has been completed and the tooth is ready to be obturated. This will reduce care provider bias.
  Assessors will be blinded to the treatment option to reduce bias during the assessment of healing.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SBO with AH Plus Bioceramic Sealer (Experimental): The teeth will be obturated using a single cone technique with AH Plus Bioceramic Sealer.
  Interventions: Device: AH Plus Bioceramic Sealer
- WVC with resin-based AH Plus Sealer (Active Comparator): The teeth will be obturated using warm vertical compaction with resin-based AH Plus Sealer.
  Interventions: Device: AH Plus Sealer (resin-based)

INTERVENTIONS:
Device: AH Plus Bioceramic Sealer — A bioactive, calcium silicate-based sealer will be used in combination with the core root canal filling material (gutta-percha). It's premixed and is dispensed in the root canal via a fine disposable syringe.
  Arms: SBO with AH Plus Bioceramic Sealer
Device: AH Plus Sealer (resin-based) — A resin-based sealer will be used in combination with the core root canal material (gutta-percha). It consists of two pastes that are mixed together in equal amounts prior to application.
  Arms: WVC with resin-based AH Plus Sealer

SUMMARY:
The goal of this clinical trial is to assess the efficacy and outcome of sealer-based obturation (SBO) using a new calcium silicate sealer in comparison with warm vertical compaction (WVC) using a resin-based sealer, which is the current gold standard.

DETAILED DESCRIPTION:
Calcium silicate sealers are used in endodontics because of their biocompatibility, bioactivity, and their ability to form a hydroxyapatite-mediated interfacial bond with root canal dentine. Although in vitro and retrospective clinical studies have reported promising findings, there remains a lack of prospective, well-controlled trials evaluating their clinical and radiographic performance.

Aims and Objectives:

1. To compare the clinical outcome of single-cone bioceramic obturation (SBO) with warm vertical compaction (WVC) in primary root canal treatment.
2. To compare the radiographic outcome of SBO and WVC using periapical (PA) radiographs and cone-beam computed tomography (CBCT).

Materials and Methods:

Patients referred for primary root canal treatment of molar teeth at Jaber Al-Ahmed Dental Center who fulfil the inclusion and exclusion criteria will be invited to participate. Written informed consent will be obtained from all participants.

Preoperative PA radiographs and CBCT scans will be taken. After completion of root canal instrumentation, participants will be randomly allocated to either Group A: SBO or Group B: WVC. Participants will be blinded to the obturation technique. Allocation will remain concealed until canals are ready for obturation, at which time the treating clinician will be informed of the assigned method.

All teeth will receive definitive restorations following obturation. Participants will be recalled at 12 months for clinical and radiographic evaluation using PA radiographs and CBCT, and will subsequently be followed annually for up to 4 years.

The study will conform to the CONSORT statement and will be conducted in accordance with the Declaration of Helsinki. Ethical approval has been granted by the local health authority (ID: 2291).

Statistical and Analytical Plan:

Sample size estimation for the primary healing outcome was performed using PASS (NCSS, Kaysville, UT, USA). Burns et al. (2022) reported pooled healing rates of approximately 92-93% under loose criteria and 82% under strict criteria in primary NSRCT, indicating that reductions on the order of 10-12 percentage points are clinically meaningful. Based on these data, an absolute 12% difference (0.99 vs 0.87) was considered clinically important.

Using a two-sided test comparing two independent proportions, with 80% power and 5% significance level, detecting this 12% absolute difference required 108 teeth (54 per group). Accounting for a 20% anticipated loss to follow-up, the required sample size is 136 teeth (68 per group).

Healing at 12 months will serve as the dependent variable in logistic regression models. Predictor variables will include age, sex, preoperative status, presence of apical periodontitis, preoperative pain, patency, apical preparation size, root filling quality, and sealer type. Two-way interactions will be assessed. Analyses will follow the intention-to-treat principle.

Null Hypothesis:

H₀: There is no difference between SBO and WVC in clinical or radiographic healing outcomes at 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be 18-65 years of age at the time of recruitment
* Participants must have a classification of I or II on the American Society of Anesthesiologists (ASA) physical status classification system
* Participants must not have known allergies to any materials used in the study
* Participants must agree to participate in the study by signing a consent form
* Participants must have good oral hygiene
* Maxillary and mandibular permanent molar teeth that require primary root canal treatment will be included
* The teeth must be restorable and have fully formed roots with no advanced periodontal disease

Exclusion Criteria:

* ASA classification of III or more
* Pregnant or breastfeeding women
* Patients who are unable to give consent
* Patients who have advanced periodontal disease or teeth with more than 5mm probing
* Anterior, premolar and third molar teeth
* Teeth whose apices were over-enlarged at the time of pulp extirpation
* Teeth with broken instruments
* Teeth with blocked or non-negotiable canals
* Teeth with iatrogenic perforations
* Teeth with incomplete root formation
* Teeth with internal or external root resorption
* Teeth that have a poor restorative prognosis
* Teeth that require posts or extensive prosthetic rehabilitation
* Teeth with cracks
* Teeth that have been previously root-filled

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 136 (Estimated)
Dates: Start 2023-08-07 (Actual); Primary Completion 2026-01-29 (Estimated); Study Completion 2027-01-29 (Estimated)

PRIMARY OUTCOMES:
Assessment of radiographic healing with cone beam computed tomography (CBCT) scans using Estrela's PAI (periapical index) | Change from baseline periapical lesion size at 12 months
  Estrela's PAI based on CBCT will be used in logistic regression models with different predictor variables.
Assessment of clinical outcome by assessing the resolution/persistence/development of clinical signs and symptoms | Change from baseline at 12 months
  The examiner will label the teeth as having a normal clinical outcome (absence of pain, swelling and other symptoms, no sinus tract, no loss of function) or showing signs and symptoms clinical outcome (the tooth is associated with signs and/or symptoms of infection).

CONTACTS AND LOCATIONS:
Locations (1):
- Jaber Al-Ahmed Dental Center, Janūb as Surrah, Hawalli Governate, Kuwait

IPD SHARING:
Plan to Share IPD: No